CLINICAL TRIAL: NCT04723784
Title: Http://Talionis.Citic.Udc.es
Brief Title: AssessMent and Counseling to Get the Best Efficiency and Effectiveness of the Assistive TeCHnology
Acronym: MATCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The project has finished and the technological developments have been created
Sponsor: Universidade da Coruña (Other)
Collaborators: University of Alcala (Other); University of Seville (Other)
Responsible Party: Principal Investigator, Thais Pousada, PhD Professor, Universidade da Coruña
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020/597
Record Dates: First submitted 2021-01-12; First posted 2021-01-26 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Disability Physical; Disability, Learning; Disabling Disease
Keywords: Assistive technology; outcome measures; robotics; Artificial Inteligence
MeSH Terms: conditions — Learning Disabilities | interventions — Methods; Outcome Assessment, Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Person with disability (Experimental): * Initial assessment.
  * Implementation of AT in the daily life of participants
  * Application of outcome measures and analysis of the data
  Interventions: Other: Initial Assessment; Other: Implementation of assistive technology in the daily life of participants; Other: Application of outcome measures

INTERVENTIONS:
Other: Initial Assessment — In this phase the evaluation of the participants will be done, with the application of the instrument presented in outcome measures' section. According to the age of the person, specific questionnaires will be used to gather information more concrete about the skills for mobility. This assessment will allow determining the specific needs, demands and capabilities of participants. The assessment process will be done by professionals of research groups in rooms of collaborators centers.
  Other Names: Assessment of participants
Other: Implementation of assistive technology in the daily life of participants — The professionals of collaborator centers, supported by the research groups, will carry on the training in the use of AT by the participants, facilitating its incorporation during the performance of activities of daily living.
  Other Names: Intervention with AT
Other: Application of outcome measures — After the process of implementation of AT (the next 2 and 6 months), members of the research group and the professionals of collaborators centers will apply the measurement instruments to determine the possible improvements in the level of functional independence (FIM scale) of people with disabilities, the impact that the AT has had on their lifes (PIADS scale) and the level of matching between person and AT (ATD PA - MPT model).
  Other Names: Outcome measures

SUMMARY:
The best match between any person with disability and the assistive technology (AT) only can be gotten through a complete assessment and a monitoring of the needs, abilities, priorities, difficult and limitations that he/she finds in his/her life. Without this analysis, may be the risk that the AT doesn't adapt to the expectation of the person. Like this, the user, in few time, could abandon the AT device, with the unnecessary spends of resources. Therefore, is important that any project focused in the development of new innovating AT for people with disabilities includes the perspective of outcome measures as an important phase of the research. In this sense, the incorporation of the assessment, implementation process and outcome measures is vital to get the transferability during the whole project and to get the general perspective from the final user.

The protocol presents a project that aims to improve the independence, participation and functional mobility of people with disabilities.

The sample is formed by people with disabilities that will participate from the first stage of the process, with an initial assessment of their abilities and needs, a complete implication during the test of technology, and in the final application of outcome measures instruments.

Only with this perspective and active participation of the users is possible to carry on a user-centered approach. That fact will allow to define and to generate technological solutions that really adjust to the expectations, needs and priorities of the people with disabilities, avoiding that the AT be abandoned, with the consequent health and social spending.

DETAILED DESCRIPTION:
The present document is the description of a Subproject of a global and complete coordinated Project, in which are participants the University of A Coruña, the University of Alcalá de Henares and the University of Sevilla, and its title is "Artificial Intelligence and Robotic Assistive Technology devices for Disabled People" (AIR4DP).

The main result of the AIR4DP project consists of the implementation of assistive technology that allows to incorporate the latest advances in Artificial Intelligence to improve life quality of people with disabilities. With this target, the investigators present a coordinated project that is divided into three sub-projects, whose main goals consist of developing and evaluating the breakthrough of the proposed technology in people with functional diversity.

In this Study Protocol, the justification and the development of subproject MATCH are explained. It will be coordinated by the University of A Coruña, and its performance implies the participation of people with disabilities.

Therefore, this project is focused on the implementation of outcome measurement tools to improve the efficacy, effectiveness and real utility of the assistive technology devices (ATD) developed. On the other hand, it is also very important to assess the functional impact the ATD has on the user's participation in their social environment. For that, other measurement tools to assess functional mobility outcomes will also be also carried out during basal assessment and after 6 months of ATD implementation.

For this study protocol, the hypothesis is related to the relevance of the assessment of the interaction between the users and the AT: in order to guarantee a high match person-AT, to also get a positive psychosocial impact in the life of people with disabilities, the assessment and monitoring result two fundamental aspects.

According to this hypothesis, the research groups has fixed two main objectives for the MATCH subproject:

* To determine the psychosocial impact of AT created during the coordinated project (AIR4ALL) on the life of people with disabilities.
* To promote the best match between the user and the assistive technology used.

To complete, few secondary goals have been proposed:

* To assess the functional skills and abilities of people with disabilities, and to identify their needs to get independence in mobility and activities of daily living.
* To design and create the best technology solutions individualized for each person, meeting with the design for all principles, and promoting the involvement of the final user.
* To validate the assistive technology's solutions designed and prototyped in order to increase the levels of participation in daily activities to people with disabilities.
* To validate a protocol/model of outcome measures in the field of assistive technology to increase the efficiency and effectiveness of selecting and prescribing these products.

ELIGIBILITY:
Inclusion Criteria:

* People with recognized disability, derived by a disease or a permanent health status.
* Age between 2 and 21 years old.
* To form part of any of the collaborators' centers with the three universities.
* To have an independent functional level moderate - low (assessed by the Functional Independence Measure.
* To have functional skills - mobility domain level moderate - low (assessed by the Spanish version of Pediatric of Disability Inventory - PEDI)

Exclusion Criteria:

* To have any health status that is incompatible with the use of assistive technology designed and prototyped in the project.
* To have cognitive skills very limited, that limits to follow the instructions to good use of AT.
* Not to have adequate human supports to make use of AT.
* To have functional skills - mobility domain level low (assessed by the Spanish version of Pediatric of Disability Inventory - PEDI), with the need for maximum assistance from caregivers.

Ages: 24 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Psychosocial Impact of the assistive technology in the life of people with disability | Two months after the implementation phase
  Psychosocial impact of assistive technology scale (PIADS): This scale has three dimensions: competence, adaptability and Self-steem. Each of these dimensions can have a minimum value of -3 up to a maximum value of +3. Higher scores mean a better outcome
Psychosocial Impact of the assistive technology in the life of people with disability | Six months after the implementation phase
  Psychosocial impact of assistive technology scale (PIADS): This scale has three dimensions: competence, adaptability and Self-steem. Each of these dimensions can have a minimum value of -3 up to a maximum value of +3. Higher scores mean a better outcome

SECONDARY OUTCOMES:
Level of matching between person and technology | Two months after the implementation phase
  Assistive Technology Device Predisposition Assessment (ATD PA) - Device form
Level of matching between person and technology | Six months after the implementation phase
  Assistive Technology Device Predisposition Assessment (ATD PA) - Device form
Level of Independence in the performance for activities of daily living. | Two months after the implementation phase
  Functional Independence Measure (FIM). The lowest score of the scale is 18, the highest score is 126.
Level of Independence in the performance for activities of daily living | Six months after the implementation phase
  Functional Independence Measure (FIM): The lowest score of the scale is 18, the highest score is 126.

OTHER OUTCOMES:
Personal mobility: Capacity to stand up and start the walk | Two months after the implementation phase
  Test up & go
Personal mobility: Capacity to stand up and start the walk | two and six months after the implementation phase
  Test up & go
Personal mobility and walking during a 10-meter journey | Two months after the implementation phase
  10 meter walk test: The outcome of this measure is the time it takes the person to walk 10 meters
Personal mobility and walking during a 10-meter journey. | Two and six months after the implementation phase
  10 meter walk test. The outcome of this measure is the time it takes the person to walk 10 meters
Personal mobility and walking during a 6 minutes walking. | Two months after the implementation phase
  6 minute walk Test; The outocme of this test is the distance traveled during 6 minutes.
Personal mobility and walking during a 6 minutes walking. | Two and six months after the implementation phase
  6 minute walk Test; The outocme of this test is the distance traveled during 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Naya Fernández, PhD, Study Chair — Universidade da Coruña
Locations (4):
- Spain (4):
  - Faculty of Health Sciences. University of A Coruña, A Coruña, Galicia
  - University of Alcalá de Henares, Alcalá de Henares, Madrid
  - Faculty of Health Science, A Coruña
  - University of Sevilla, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groba B, Pousada T, Nieto L. Assistive technologies, tools and resources for the access and use of information and communication technologies by people with disabilities. Handbook of Research on Personal Autonomy Technologies and Disability Informatics. 2010.
- [Background] VVAA. Proyecto EASTIN. Red europea de información sobre las tecnologías para la discapacidad y la autonomía. Minusval. 2005;153:17-34.
- [Background] Laloma M. Ayudas técnicas y discapacidad. Madrid: Comité Español de Representantes de Personas con Discapacidad; 2005.
- [Background] Vidal García Alonso J, Prat Pastor J, Rodríguez-Porreor Miret C, Sández Lacuesta J, Vera Luna P. Libro Blanco I+D+I al servicio de las Personas con Discapacidad y las Personas Mayores. Vol. 1. Madrid: Ministerio de trabajo y asuntos sociales, Ministerio de Ciencia y tecnología; 2003.
- [Background] Scherer. Assistive technology matching device and consumer for successful rehabilitation. Washington DC: American psychological Association; 2001.
- [Background] Scherer M, Jutai J, Fuhrer M, Demers L, Deruyter F. A framework for modelling the selection of assistive technology devices (ATDs). Disabil Rehabil Assist Technol. 2007 Jan;2(1):1-8. doi: 10.1080/17483100600845414. PMID 19263548
- [Background] Pousada Garcia T, Groba Gonzalez B, Nieto Rivero L, Pereira Loureiro J, Diez Villoria E, Pazos Sierra A. Exploring the Psychosocial Impact of Wheelchair and Contextual Factors on Quality of Life of People with Neuromuscular Disorders. Assist Technol. 2015 Winter;27(4):246-56. doi: 10.1080/10400435.2015.1045996. PMID 26186427
- [Background] DeRuyter. The importance of outcome measures for assistive tehcnology service delivery systems. Technol Disabil. 1997;6:89-104.
- [Background] World Health Organization. Global priority research agenda for improving access to high-quality affordable assistive technology The Initiative [Internet]. Geneva; 2017 [cited 2017 Jul 18]. Available from: http://apps.who.int/iris/bitstream/10665/254660/1/WHO-EMP-IAU-2017.02-eng.pdf?ua=1
- [Background] Fuhrer MJ, Jutai JW, Scherer MJ, DeRuyter F. A framework for the conceptual modelling of assistive technology device outcomes. Disabil Rehabil. 2003 Nov 18;25(22):1243-51. doi: 10.1080/09638280310001596207. PMID 14617441
- [Background] Smith RO, Rust KL, Jansen C, & Seitz J. ATOMS Project technical report - The ICF in the context of assistive technology (AT) interventions and outcomes [Internet]. Vol. 2010. 2006. Available from: http://www.r2d2.uwm.edu/atoms/archive/icf.html.
- [Background] Jimenez Arberas E. "Impacto psicosocial de los productos y tecnologías de apoyo para la comunicación en personas con discapacidad auditiva y personas sordas [Internet]. University of Salamanca; 2016. Available from: http://sid.usal.es/idocs/F8/FDO27380/JimenezArberas.pdf
- [Background] Pousada Garcia T. Impacto psicosocial de la silla de ruedas en la vida de las personas con enfermerades neuromusculares. [A Coruña]: Universidade da Coruña; 2011.
- [Background] Groba B, Pousada T, Nieto L. Assistive technologies, tools and resources for the access and use of information and communication technologies by people with disabilities. Assistive Technologies: Concepts, Methodologies, Tools, and Applications. 2013.
- [Background] Pousada T, Groba B, Nieto-Riveiro L, Pazos A, Diez E, Pereira J. Determining the burden of the family caregivers of people with neuromuscular diseases who use a wheelchair. Medicine (Baltimore). 2018 Jun;97(24):e11039. doi: 10.1097/MD.0000000000011039. PMID 29901600
- [Background] Pousada T, Pereira-Loureiro J, Díez E, Groba B, Nieto-Riveiro L, Pazos A. Needs, demands and reality of people with neuromuscular disorders users of wheelchair. Examines Phys Med Rehabil [Internet]. 2017 Nov 13 [cited 2019 Jul 15];1(1). Available from: https://ruc.udc.es/dspace/handle/2183/20294
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Mylius CF, Paap D, Takken T. Reference value for the 6-minute walk test in children and adolescents: a systematic review. Expert Rev Respir Med. 2016 Dec;10(12):1335-1352. doi: 10.1080/17476348.2016.1258305. Epub 2016 Nov 21. PMID 27817221
- [Background] Peters DM, Fritz SL, Krotish DE. Assessing the reliability and validity of a shorter walk test compared with the 10-Meter Walk Test for measurements of gait speed in healthy, older adults. J Geriatr Phys Ther. 2013 Jan-Mar;36(1):24-30. doi: 10.1519/JPT.0b013e318248e20d. PMID 22415358
- [Background] Garcia C. Adaptación transcultural y validación de la versión en español de la Pediatric Balance Scale. Universidad de Extremadura; 2017.
- [Background] Uniform Data System for Medical. Functional Independence Measure, version 5.1. New York: Buffalo General Hospital; 1997.
- [Background] Martinez-Martin P, Fernandez-Mayoralas G, Frades-Payo B, Rojo-Perez F, Petidier R, Rodriguez-Rodriguez V, Forjaz MJ, Prieto-Flores ME, de Pedro Cuesta J. [Validation of the functional independence scale]. Gac Sanit. 2009 Jan-Feb;23(1):49-54. doi: 10.1016/j.gaceta.2008.06.007. Epub 2009 Jan 9. Spanish. PMID 19231723
- [Derived] Pousada Garcia T, Groba Gonzalez B, Nieto-Riveiro L, Canosa Dominguez N, Maldonado-Bascon S, Lopez-Sastre RJ, Pacheco DaCosta S, Gonzalez-Gomez I, Molina-Cantero AJ, Pereira Loureiro J. Assessment and counseling to get the best efficiency and effectiveness of the assistive technology (MATCH): Study protocol. PLoS One. 2022 Mar 16;17(3):e0265466. doi: 10.1371/journal.pone.0265466. eCollection 2022. PMID 35294488

DOCUMENTS (1):
  • Study Protocol (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT04723784/Prot_000.pdf